CLINICAL TRIAL: NCT04511676
Title: The Study of Pharmacokinetics of Levetiracetam in Patients Undergoing Intermittent Hemodialysis
Status: Completed | Type: Observational
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Other Study IDs: LEV-HD
Record Dates: First submitted 2020-07-31; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Seizures
Keywords: Levetiracetam; Pharmacokinetics; Hemodialysis
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Levetiracetam (LEV) is one of second-generation antiepileptic drugs that has been used to treat partial and generalized epilepsy. LEV is eliminated from the systemic circulation by renal excretion. Therefore, patients with renal impairment may experience a reduced drug excretion and increased adverse drug reactions. Moreover, patients with end-stage renal disease who need dialysis may experience low serum LEV concentration because of drug loss via dialysis. LEV loss via dialysis can cause low serum level of LEV that insufficient for seizure control. The present study was aimed to evaluate pharmacokinetics of LEV in patients undergoing 4 hour-intermittent hemodialysis (IHD). The results of the study may benefit to determine the appropriate LEV initial dose and supplemental dose for patients undergoing IHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were at least 18 years old.
2. Patients who were diagnosed with seizure.
3. Patients who were undergoing intermittent hemodialysis and were treated with intravenous Levetiracetam not less than 2 days

Exclusion Criteria:

1. Patients who were pregnant or lactating
2. Patients who were treated with intravenous Levetiracetam more than once a day
3. Patients who were undergoing sustained low efficiency dialysis (SLED)
4. Patients who have intermittent dialysis duration less than 3 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to Phramongkutklao Hospital as inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Levetiracetam | Immediately before an initiation of an intermittent hemodialysis session
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | 1 hour after an initiation of an intermittent hemodialysis session
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | 2 hour after an initiation of an intermittent hemodialysis session
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | 3 hour after an initiation of an intermittent hemodialysis session
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | 4 hour after an initiation of an intermittent hemodialysis session
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | Before an administration of Levetiracetam post-hemodialysis supplemental dose
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day
Plasma concentration of Levetiracetam | 1 hour after finishing an administration of Levetiracetam post-hemodialysis supplemental dose
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on dialysis day

SECONDARY OUTCOMES:
Plasma concentration of Levetiracetam | Immediately before Levetiracetam administration
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on non-dialysis day.
Plasma concentration of Levetiracetam | 1 hour after finishing Levetiracetam administration
  Measured Levetiracetam plasma concentration (mcg/mL) of the subjects on non-dialysis day.
Number of participants with adverse drug reactions from Levetiracetam | From the first day that participants were included to the study and treated with Levetiracetam until the date of the last point of serum Levetiracetam sampling, assessed up to 3 days
  Observed signs and symptoms of Levetiracetam adverse drug reactions after participants were administered with Levetiracetam.

CONTACTS AND LOCATIONS:
Overall Officials: Pasiri Sithinamsuwan, MD, Study Chair — Pharmongkutklao Hospital and College of Medicine; Daraporn Rungprai, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Juthathip Suphanklang, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Wongsakorn Promken, B Pharm, Principal Investigator — The College of Pharmacotherapy of Thailand
Locations (1):
- Pharmongkutklao Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patsalos PN. Pharmacokinetic profile of levetiracetam: toward ideal characteristics. Pharmacol Ther. 2000 Feb;85(2):77-85. doi: 10.1016/s0163-7258(99)00052-2. PMID 10722121
- [Background] Patsalos PN. Clinical pharmacokinetics of levetiracetam. Clin Pharmacokinet. 2004;43(11):707-24. doi: 10.2165/00003088-200443110-00002. PMID 15301575
- [Background] Smetana KS, Cook AM, Bastin ML, Oyler DR. Antiepileptic dosing for critically ill adult patients receiving renal replacement therapy. J Crit Care. 2016 Dec;36:116-124. doi: 10.1016/j.jcrc.2016.06.023. Epub 2016 Jul 5. PMID 27546759
- [Background] Engelbrecht L, Grobler CJ, Rheeders M. A simple and cost-effective HPLC-UV method for the detection of levetiracetam in plasma/serum of patients with epilepsy. Biomed Chromatogr. 2017 Oct;31(10). doi: 10.1002/bmc.3969. Epub 2017 Apr 20. PMID 28294369
- [Background] Jarvie D, Mahmoud SH. Therapeutic Drug Monitoring of Levetiracetam in Select Populations. J Pharm Pharm Sci. 2018;21(1s):149s-176s. doi: 10.18433/jpps30081. PMID 30096051
- [Background] Yamamoto J, Toublanc N, Kumagai Y, Stockis A. Levetiracetam pharmacokinetics in Japanese subjects with renal impairment. Clin Drug Investig. 2014 Nov;34(11):819-28. doi: 10.1007/s40261-014-0237-7. PMID 25312351
- [Background] Shiue HJ, Taylor M, Sands KA. Comparison of Levetiracetam Dosing Regimens in End-Stage Renal Disease Patients Undergoing Intermittent Hemodialysis. Ann Pharmacother. 2017 Oct;51(10):862-865. doi: 10.1177/1060028017713294. Epub 2017 Jun 5. PMID 28582998
- [Background] Wieruszewski PM, Kashani KB, Rabinstein AA, Frazee E. Levetiracetam Pharmacokinetics in a Critically Ill Anephric Patient on Intermittent Hemodialysis. Neurocrit Care. 2018 Apr;28(2):243-246. doi: 10.1007/s12028-017-0441-4. PMID 28828726
- [Background] Company-Albir MJ, Ruiz-Ramos J, Solana Altabella A, Marques-Minana MR, Vicent C, Poveda JL. Haemodialysis significantly reduces serum levetiracetam levels inducing epileptic seizures: Case report. J Clin Pharm Ther. 2017 Dec;42(6):774-775. doi: 10.1111/jcpt.12568. Epub 2017 May 28. PMID 28555936